CLINICAL TRIAL: NCT06905353
Title: Quality of Recovery in the Post-anesthesia Care Unit - Minimal Clinically Important Difference and Correlation with Postoperative Quality of Recovery One Day After Non-cardiac Surgery
Brief Title: Quality of Recovery in the Post-anesthesia Care Unit
Acronym: MiDiQoR
Status: Not yet recruiting | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-101434-BO-ff
Record Dates: First submitted 2025-03-25; First posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Postoperative Quality of Recovery; Postoperative Quality of Recovery in the Postanesthesia Care Unit
Keywords: postoperative care; patient-reported outcome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- MCID: patients that will answer the QoR-PACU2 twice with anchor questions to identify the minimal clinically important difference
- correlation: patients that will additionally answer the QoR-15GE before surgery and on postoperative day one

SUMMARY:
This prospective observational study aims to identify the minimal clinically important difference of the QoR-PACU2 questionnaire. In addition, this study aims to assess the correlation between self-reported quality of postoperative recovery early after surgery in the post-anesthesia care unit and postoperative recovery on the first day after surgery.

ELIGIBILITY:
Inclusion Criteria:

* elective non-cardiac surgery
* expected duration of surgery ≥60 minutes
* postoperative stay at the post-anesthesia care unit

Exclusion Criteria:

* surgery or condition requiring postoperative treatment at an intensive care unit
* inability to give informed consent/requirement of a legal guardian

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients scheduled for elective non-cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 188 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Minimal clinically important difference of QoR-PACU2 | From preoperative assessment to the day of surgery in the post-anesthesia care unit
  The minimal difference in the QoR-PACU2 scores that is relevant for the patient
correlation between quality of recovery at two time points of assessment | from the day of surgery to the first postoperative day
  The correlation between quality of recovery in the post-anesthesia care unit and quality of recovery on postoperative day one

IPD SHARING:
Plan to Share IPD: No